CLINICAL TRIAL: NCT03590119
Title: Intra-arterial Lutetium-177-dotatate for Treatment of Patients With Neuro-endocrine Tumor Liver Metastases
Acronym: LUTIA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Marnix Lam (Other)
Responsible Party: Sponsor-Investigator, Marnix Lam, Prof. dr. M.G.E.H. Lam, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL60725.041.17
Record Dates: First submitted 2018-07-03; First posted 2018-07-18 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Neuroendocrine Tumors; Liver Metastases
Keywords: LUTIA; neuroendocrine tumor; lutetium-177-dotatate; intra-arterial; liver metastases
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Intervention Model Description: This study uses a with-in subject randomization between intra-arterial treatment via the left or right hepatic artery.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-arterially treated liver lobe (Experimental): Depending on the allocation after randomization, Lu-177-dotatate will be infused in either the left or the right hepatic artery, following catheterization using the Seldinger-technique.
  Interventions: Drug: Lutetium Lu 177-DOTATATE
- 'Intravenously' treated liver lobe (Active Comparator): The lobe that is not treated intra-arterially, will act as the intravenously treated lobe, due to the first-pass effect.
  Interventions: Drug: Lutetium Lu 177-DOTATATE

INTERVENTIONS:
Drug: Lutetium Lu 177-DOTATATE — Intra-arterial infusion of Lu-177-DOTATATE
  Other Names: Lutathera

SUMMARY:
The objective is to investigate the impact of intra-arterial administration of 177Lu-dotatate on the intrahepatic biodistribution in patients with NET liver metastases. Our primary objective is to evaluate if there is a difference in post-treatment tumor-to-non-tumor (T/N) activity concentration ratio on SPECT/CT between the intra-arterial treated liver lobe and the intravenous treated liver lobe.

DETAILED DESCRIPTION:
Rationale: The majority of neuroendocrine tumor (NET) patients present with metastases, most often including liver metastases. These patients have a poorer prognosis and lower quality of life.

Currently, intravenous administered somatostatin-bound radionuclides (177Lu-dotatate) have shown to improve tumor response rates and progression free survival (PFS). Despite of the increased tumor response rate and PFS, liver metastases still remain the major cause of morbidity and mortality in these patients. Patients with liver metastases have a worse outcome in terms of overall survival after treatment with 177Lu-dotatate compared to patients with limited or no liver metastases.

Objective: to investigate the impact of intra-arterial (IA) administration of 177Lu-dotatate on the intrahepatic biodistribution in patients with NET liver metastases. Our primary objective is to evaluate if there is a difference in post-treatment tumor-to-non-tumor (T/N) activity concentration ratio on SPECT/CT between the intra-arterial treated liver lobe and the intravenous treated liver lobe.

Study design: Multicenter, interventional, block randomized, phase 2 clinical trial. We use a within-subject controlled design where the administration of 177Lu-dotatate is randomized between the right or left hepatic artery. Selective IA administration of 177Lu-dotatate allows for intra-patient comparison between IA administration (one lobe) versus IV 'administration' (the other lobe). The contralateral liver lobe and the rest of the body receive treatment by second pass IV route.

Study population: 26 patients with NET liver metastases (> 18 years old). Intervention: Treatment will be randomized between selective right or left hepatic artery administration of 177Lu-dotatate (Four administrations of 7.4 GBq; each via the same randomly allocated hepatic artery during angiography).

Main study parameters/endpoints: To assess if there is a difference in post-treatment tumor-to-non-tumor (T/N) activity concentration ratio on SPECT/CT between the intra-arterial treated liver lobe and the intravenous treated liver lobe. The T/N activity concentration will be measured on SPECT/CT. The primary endpoint will be assessed after the first treatment cycle. The T/N activity ratios of the second, third, and final treatment cycle will be assessed as secondary endpoint. Tumor response, toxicity, extrahepatic uptake and kidney uptake are secondary endpoints. Intra- and inter-patient differences will be studied.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: As with the standard IV treatment with 177Lu-dotatate, the treatment consists of four cycles. During each cycle, patients will be admitted for 1 night and undergo physical examination, laboratory examination, angiography with administration of the treatment dose, and post-treatment imaging. Risks include standard complication risks related to angiography (bleeding or infection). No additional risks with relation to the treatment itself are expected compared to the standard IV treatment (nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have given written informed consent.
* Female or male aged 18 years and over.
* Inoperable histologically proven neuro-endocrine tumor with indication for 177Lu-dotatate at enrollment time.
* Well-differentiated neuro-endocrine tumor with a Ki67-index ≤20% and a mitotic count of ≤20.
* Confirmed presence of somatostatin receptors on target lesions, based on somatostatin receptor imaging.
* Life expectancy of 6 months or longer.
* Eastern Cooperative Oncology Group (ECOG) performance score 0-1.
* Hepatic metastases with at least one lesion ≥3 cm on cross sectional imaging in both the right and left liver lobe (i.e. left and right lobes are based on the hepatic arterial perfusion territory).
* Presence of excessive liver metastases, defined as >25% tumor load, with or without extrahepatic metastases.
* Patients must have clinical or radiological progressive disease.
* Negative pregnancy test for women of childbearing potential.

Exclusion Criteria:

* Any previous radioembolization, chemoembolization, or bland embolization, at any time, or surgery or radiofrequency ablation (or other ablative therapies) within 12 weeks prior to randomization in the study.
* Prior external beam radiation therapy to the liver.
* Interferons, Everolimus (mTOR-inhibitors) or other systemic therapies within 4 weeks prior to randomization in the study.
* Any patient receiving treatment with short-acting Octreotide, which cannot be interrupted for 24 hours before and 24 hours after the administration of 177Lu-dotatate, or any patient receiving treatment with Octreotide LAR, which cannot be interrupted for at least 4 weeks before the administration of 177Lu-dotatate, unless the tumor uptake on target lesions observed by imaging during continued Octreotide LAR treatment is higher than normal liver uptake.
* Any unresolved toxicity greater than National Cancer Institute (NCI), Common Terminology Criteria for Adverse Events (CTCAE version 4.03) grade 2 from previous anti-cancer therapy.
* Serum bilirubin > Upper Limit of Normal (ULN), serum albumin <3.0 g/dL.
* Glomerular filtration rate <50 ml/min.
* Hb <5.5 mmol/L; leucocytes <3.0x109/L; platelets <100x109/L (at baseline; 75x109/L is sufficient for cycles 2-4).
* Uncontrolled congestive heart failure (NYHA II, III, IV).
* Uncontrolled diabetes mellitus.
* Patients suffering from diseases with an increased chance of liver toxicity.
* Patients suffering from psychic disorders that make a comprehensive judgement impossible, such as psychosis, hallucinations and/or depression. Patients who are declared incompetent.
* Previous enrolment in the present study or previous treatment with 177Lu-dotatate.
* Female patients who are not using an acceptable method of contraception (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal ligation) OR are less than 1 year postmenopausal or surgically sterile during their participation in this study (from the time they sign the consent form) to prevent pregnancy.
* Male patients who are not surgically sterile or do not use an acceptable method of contraception during their participation in this study (from the time they sign the consent form) to prevent pregnancy in a partner.
* Body weight over 150 kg.
* Current spontaneous urinary incontinence.
* Severe allergy for i.v. contrast (Visipaque®), used for CT evaluation and treatment angiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
The difference in post-treatment tumor-to-non-tumor (T/N) activity concentration ratio on SPECT/CT between the intra-arterial treated liver lobe and the intravenous treated liver lobe. | 24 hours
  To assess if there is a difference in post-treatment tumor-to-non-tumor (T/N) activity concentration ratio on SPECT/CT between the intra-arterial treated liver lobe and the intravenous treated liver lobe. The T/N activity concentration will be measured on SPECT/CT. The primary endpoint will be assessed after the first treatment cycle. For each liver lobe up to three tumors (i.e. all >3 cm) will be selected based on size (i.e. the largest lesions without central necrosis). The weighted average activity per voxel of these lesions will be divided by the normal liver tissue mean activity per voxel (i.e. a VOI with 3 cm diameter will be placed in the normal liver tissue) to calculate the T/N ratio. The T/N activity ratios of the second, third, and final treatment cycle will be assessed as secondary endpoint. Intra- and inter-patient differences will be studied.

SECONDARY OUTCOMES:
The difference in absolute values of mean tumor and healthy liver absorbed dose on post-treatment SPECT/CT between the intra-arterial treated liver lobe and the intravenous treated liver lobe | 24 hours
  Difference in absolute values of mean tumor and healthy liver absorbed dose (in Gy) on post-treatment SPECT/CT between the intra-arterial treated liver lobe and the intravenous treated liver lobe: Dosimetry will be performed to measure mean tumor and healthy liver absorbed dose. Dosimetry will be performed on post-treatment SPECT/CT, which is performed 24 hours after administration of 177Lu-dotatate. The absolute absorbed dose in the IA treated liver lobe will be compared to the IV treated lobe.
The difference in post-treatment tumor response between the intra-arterial treated liver lobe and the intravenous treated liver lobe | 3 and 6 months
  -Difference in post-treatment tumor response between the intra-arterial treated liver lobe and the intravenous treated liver lobe: The tumors are measured on CT and scored according to the Southwest Oncology Group (SWOG) solid tumor response criteria, RECIST 1.1, and mRECIST criteria. Scoring systems will be applied on the patient and liver level, separately.
  Because the eventual maximal shrinkage of the tumors may take months after completion of the therapy, we added the tumor response class 'minimal response (MR)', pertaining to a decrease in summed squares of tumor diameter more than 25% but less than 50%.
The dose-response relation between tumor absorbed dose and post-treatment tumor response | 3 and 6 months
  To assess if there is a dose-response relation between tumor absorbed dose and post-treatment tumor response: The tumor absorbed dose in both the IA and IV treated liver lobe will be calculated based on SPECT/CT as mentioned above. Tumor response will be measured on post-treatment follow-up imaging. With these parameters, a possible dose-response relation will be evaluated.
Toxicity and how toxicity is compared to historical controls | 6 months
  To assess safety and toxicity according to the common toxicity criteria on adverse events (CTCAE) version 4.03. The grade of toxicity refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE. Especially myelo-toxicity, renal toxicity and hepatic toxicity will be evaluated.
Sufficient uptake of 177Lu-dotatate in extrahepatic lesions | 24 hours
  To assess if there is sufficient uptake of 177Lu-dotatate in extrahepatic lesions (comparison will be made with historical data): The 177Lu-dotatate uptake of the extrahepatic lesions (e.g. pancreas, intestine) will be calculated on post-treatment SPECT/CT. These results will be compared to historical data in order to evaluate if these extrahepatic tumor sites show sufficient uptake.
Sufficient uptake of 177Lu-dotatate in the contralateral lobe, compared to historical controls | 24 hours
  To assess if there is sufficient uptake of 177Lu-dotatate in the contralateral lobe (comparison will be made with historical data): The 177Lu-dotatate uptake of the contralateral lobe will be calculated on post-treatment SPECT/CT. These results will be compared to historical data in order to evaluate if the other lobe shows sufficient uptake.
The difference in kidney uptake of 177Lu-dotatate between the IA treated patients and historical controls | 24 hours
  To assess if there is a difference in kidney uptake of 177Lu-dotate between the IA treated patients and historical controls: Kidney uptake will be calculated on post-treatment SPECT/CT and compared to historical controls in order to assess differences in uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Marnix GEH Lam, MD PhD, Principal Investigator — UMC Utrecht
Locations (3):
- Netherlands (3):
  - Antoni van Leeuwenhoek Cancer Institute, Amsterdam
  - Erasmus MC, Rotterdam
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ebbers SC, Braat AJAT, Moelker A, Stokkel MPM, Lam MGEH, Barentsz MW. Intra-arterial versus standard intravenous administration of lutetium-177-DOTA-octreotate in patients with NET liver metastases: study protocol for a multicenter, randomized controlled trial (LUTIA trial). Trials. 2020 Feb 5;21(1):141. doi: 10.1186/s13063-019-3888-0. PMID 32024533